CLINICAL TRIAL: NCT06117072
Title: Which Is More Effective in Hypertension?: Salt-Free Diet vs. DASH Diet
Brief Title: Hypertension DASH Diet and Salt Free Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Aslı Gizem Çapar, Principal Investigator, Nuh Naci Yazgan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NuhNaciYU
Record Dates: First submitted 2023-10-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Hypertension; Nutritional Status; Diet, Healthy; Blood Pressure; Salt; Deficit (or Low)
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This randomized controlled intervention study aimed to compare the effects of a Dietary Approaches to Stop Hypertension (DASH) diet and a salt-free diet on blood pressure in hypertension patients. Methods: This study was conducted with 60 patients with primary hypertension. One group (n=30) was given an individualized DASH diet, the other group was given a salt-free diet (n=30), and the participants were followed for two months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dash diet group, salt free diet (Experimental): This randomized controlled intervention study aimed to compare the effects of a Dietary Approaches to Stop Hypertension (DASH) diet and a salt-free diet on blood pressure in hypertension patients. Methods: This study was conducted with 60 patients with primary hypertension. One group (n=30) was given an individualized DASH diet, the other group was given a salt-free diet (n=30), and the participants were followed for two months.
  Interventions: Other: diet plan

INTERVENTIONS:
Other: diet plan — One group (n = 30) received the DASH diet and the other group received a salt-free diet (n = 30) and was followed for 2 months

SUMMARY:
Background: In the management of hypertension lifestyle changes are recommended along with pharmacological treatment.

Aims: This randomized controlled intervention study aimed to compare the effects of a Dietary Approaches to Stop Hypertension (DASH) diet and a salt-free diet on blood pressure in hypertension patients. Methods: This study was conducted with 60 patients with primary hypertension. One group (n=30) was given an individualized DASH diet, the other group was given a salt-free diet (n=30), and the participants were followed for two months. The patients' blood pressures were monitored daily throughout the study, and their biochemical parameters were monitored at the beginning of the study, in the first and second months.

DETAILED DESCRIPTION:
This study, which was planned as a randomized controlled intervention study, was conducted to compare the effects of the Dietary Approaches to Stop Hypertension (DASH) and salt-free diet on blood pressure in patients with hypertension. The study was complited with the participation of 60 hypertensive individuals (46 females, 14 males) who applied to between July 2019 and March 2020. Patients with hypertension who were living in Kayseri province, at least elementary school graduate, in the 20-65 age group, able to communicate with the researcher face to face and by phone, diagnosed with hypertension at least 4 weeks ago, and whose medication did not change were included in the study. One group (n = 30) received the DASH diet and the other group received a salt-free diet (n = 30) and was followed for 2 months. Research data was repeated during application with the face-to-face interview method. Research data was collected through a questionnaire containing questions about the sociodemographic characteristics, nutritional habits, chronic diseases, and medications of the individuals. Anthropometric measurements of the patients were made and blood and urine samples were taken. Food consumption frequency was noted, DASH diet compliance scale and International Physical Activity Questionnaire (IPAQ) short form were applied.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension at least four weeks prior and had not changed their drug regimen in the previous four weeks
* 20-65 age group
* At least primary school graduate
* Able to express himself verbally
* Volunteer to participate in the dietary intervention
* Able to communicate with the researcher face to face and by phone

Exclusion Criteria:

* Those with chronic diseases other than cardiovascular diseases (such as Type II diabetes, kidney disease, cancer disease)
* Using alcohol or smoking

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
comparison of blood pressure measurements | two months
  blood pressure (mmHg)
comparison of anthropometric measurements | two months
  body weight (kg)
comparison of anthropometric measurements | two months
  height (m)
comparison of anthropometric measurements | two months
  body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Asli Gizem Çapar, Kayseri, Kayseri̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
data can be shared if necessary